CLINICAL TRIAL: NCT02462174
Title: Caudal Epidural Block Versus Topical Ketamine Application for Postoperative Pain Relief After Elective Inguinal Herniotomy
Brief Title: Topical Ketamine Versus Caudal Ketamine for Postoperative Analgesia in Children Undergoing Inguinal Herniotomy
Acronym: TKversusCK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, assistant professor anesthesia and intensive care department/ faculty of medicine/ Assiut university/ Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/ NF
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
Keywords: anesthesia; analgesia; caudal; ketamine; bupivacaine
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical ketamine and topical bupivacaine (Active Comparator): 0.5 mg/ kg ketamine in 0.3 ml/kg bupivacaine 0.25% (maximum volume = 20 ml) administered directly around the spermatic cord in the wound after end of surgery and before closure of the wound.
  Interventions: Drug: Ketamine; Drug: Bupivacaine
- Caudal ketamine and caudal bupivacaine (Active Comparator): 0.5 mg/ kg ketamine in 1 ml/kg bupivacaine 0.25% (maximum volume = 20 ml) administered by caudal epidural route after anesthesia and before the start of surgery.
  Interventions: Drug: Ketamine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/ kg ketamine with bupivacaine by caudal route after anesthesia and before start of surgery.
  Other Names: Katalar
  Arms: Topical ketamine and topical bupivacaine
Drug: Ketamine — 0.5 mg/ kg ketamine with bupivacaine will be sprayed around the spermatic cord before wound closure.
  Other Names: Katalar
  Arms: Caudal ketamine and caudal bupivacaine
Drug: Bupivacaine — 1 ml/kg bupivacaine 0.25% (maximum volume = 20 ml) by caudal route
  Other Names: bucaine
  Arms: Topical ketamine and topical bupivacaine
Drug: Bupivacaine — 0.3 ml/kg bupivacaine 0.25% will be sprayed around the spermatic cord before wound closure
  Other Names: bucaine
  Arms: Caudal ketamine and caudal bupivacaine

SUMMARY:
To find alternatives to caudal analgesia that could be more safe and effective and to demonstrate the analgesic efficacy of topical ketamine.

DETAILED DESCRIPTION:
The most commonly performed inguinal surgeries in children include inguinal hernia repair with or without orchidopexy (orchiopexy). Eighty children aged 6 months to 6 yr of ASA physical status I or II, undergoing elective unilateral inguinal herniotomy will be included. In caudal group, patients will receive a mixture of 0.5 mg/ kg ketamine in 1 ml/kg bupivacaine 0.25% (maximum volume = 20 ml) by caudal route after anesthesia and before start of surgery. In topical group, at the end of the procedure, after identification and ligation of the hernial sac, a mixture of 0.5 mg/ kg ketamine in 0.3 ml/kg bupivacaine 0.25% will be sprayed around the spermatic cord and upon the ilioinguinal nerve in a fan shaped manner by the surgeon. The primary outcome measure will be the time to first request for analgesia. Secondary outcome measures will include the number of analgesic doses required in the first 24 h postoperative, pain scores, sensory and motor block, agitation scores, parent satisfaction and adverse effects in the first 48h postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. age (6 months to 6 years)
2. ASA physical status I or II.
3. Operation: elective unilateral inguinal herniotomy.

Exclusion Criteria:

1. A history of developmental delay or mental retardation,
2. Known or suspected coagulopathy,
3. Known allergy to any local anaesthetic,
4. Known congenital anomaly of the spine or signs of spinal anomaly,
5. Infection at the sacral region.

Ages: 6 Months to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
time to first request for postoperative analgesia | 48 hours postoperative
  time in hours from admission to PACU till first request for analgesia

SECONDARY OUTCOMES:
total consumption of postoperative analgesics | 48 hours postoperative
  the amount of analgesic drugs in mg given in the first 48h postoperative
The Children's Hospital of Eastern Ontario Pain Scale (CHEOPS, 0-10) pain score | 180 minutes postoperative
Faces Legs Activity Cry Consolability tool (FLACC, 0-10). | 180 minutes postoperative.
the agitation score (0= child is asleep, 1= awake/calm, 2= irritable/ consolable cry, 3=inconsolable cry, 4= the child is agitating and thrashing and restlessness). | 60 minutes postoperative
parent's satisfaction on a four-point Likert scale (1, excellent; 2, good; 3, fair; 4, poor). | 48 hours postoperative
  the score will be recorded once at the end of the study
noninvasive blood pressure | Intra-operative
heart rate | Intra-operative
Verbal Numeric Rating Scale (VNRS) | 48 hours postoperative
  the pain score will be assessed at frequent intervals in the 1st 48 h postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt